CLINICAL TRIAL: NCT05629988
Title: Observational Study of Repeat Immunoadsorption (RIA) in Post Covid ME/CFS Patients With Elevated ß2 Adrenergic Receptor Autoantibodies
Brief Title: Repeat Immunoadsorption Post Covid ME/CFS
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Carmen Scheibenbogen, Director of the Institute for Medical Immunology, Charite University, Berlin, Germany
Other Study IDs: IAINPCS; 01EP2201 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2022-11-14; First posted 2022-11-29 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Post-COVID ME/CFS
Keywords: Post-COVID Syndrome; Long COVID; Chronic Fatigue Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: IA with TheraSorb ® column — IA cycle is 5 days, repeat cycles will be given to responders at months 3 and 6

SUMMARY:
The evidence for an autoimmune etiology in postinfectious myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS) is growing. The investigators observed in a not yet published study that in ME/CFS triggered by COVID, similar to ME/CFS after other infections, there is a close correlation of ß2 adrenergic receptor (ß2R) autoantibodies with symptom severity.

Immunoadsorption (IA) to remove autoantibodies has been used successfully in many autoantibody-mediated diseases. The investigators have already performed two proof of concept studies of IA in postinfectious ME/CFS with elevated ß2R antibodies, which resulted in improvement in most patients. This observational study aims to assess symptom outcome and functional ability in 20 patients with Post-COVID Syndrome (PCS) meeting ME/CFS diagnostic criteria with elevated ß2R antibodies undergoing antibody depletion by IA. The study will be conducted as a non-interventional observational study. IA with Miltenyi's TheraSorb® column in PCS will be performed in the approved use. Patients who have symptom improvement after the 1st IA will receive two additional IAs at 3 and 6 months, which will also be documented.

The results of this observational study will provide the basis for a randomized controlled clinical trial (RCT) combining IA with B-cell depletion therapy preferentially with Obinutuzumab.

DETAILED DESCRIPTION:
Studies indicate an overlap between post-COVID syndrome (PCS) and ME/CFS (Kedor et al., 2022). Post-infectious ME/CFS (ICD-10 code G93.3) is a complex and severely disabling disease with no approved treatment and thus, a very high medical need. Following an acute infection, patients suffer from severe central and muscle fatigue, chronic pain, cognitive impairment, and immune and autonomic dysfunction. The key symptom of ME/CFS is exertion intolerance with minor exertion resulting in symptom aggravation, also called post-exertional malaise (PEM), lasting until the next day up to weeks.

Various pathogens are known to induce post-infectious ME/CFS, including the Epstein-Barr virus and SARS-CoV-2 (Sotzny, 2018). The investigators' ongoing Charité PA-COVID study (Berlin prospective COVID-19 patient cohort) and other reports show that SARS-CoV-2 triggers ME/CFS in a subset of mostly younger patients without preexisting comorbidities (Kedor et al., 2022). Due to the rapid increase of COVID-19 incidence worldwide, the prevalence of post-COVID-19 ME/CFS will likely be a substantial problem for health care and society.

The evidence for an autoimmune etiology in post-infectious ME/CFS is growing (reviewed in Sotzny et al., 2018). Also, COVID-19 is a disease with a high risk for autoimmunity and developing ME/CFS due to the infection of many different cell types and the severity of immune activation. There is evidence from several studies from the investigators and other groups that natural regulatory autoantibodies targeting G protein-coupled receptors (GPCR) are involved in the pathogenesis of various autoimmune diseases. The investigators and others described enhanced levels and dysfunction of ß2R autoantibodies in ME/CFS and their correlation with the severity of key clinical symptoms (Freitag et al., 2021). The investigators' working hypothesis is that GPCR-specific autoantibodies with altered binding affinity or epitope specificity lead to immune dysregulation and autonomous dysfunction, and play a significant role in the pathomechanism of ME/CFS (Wirth et al., 2020). The investigators observed -- in a not yet published study -- a close correlation of ß2R antibodies with symptom severity in ME/CFS after COVID, similar to ME/CFS after other infections (Freitag et al., 2021). Two small proof-of-concept studies with immunoadsorption (IA) in patients with ME/CFS after other infections have shown improvements in symptoms in most patients (Scheibenbogen et al., 2018; Toelle et al., 2020).

In this observational non-controlled trial, PCS ME/CFS patients who receive IA will be evaluated for clinical efficacy, a decrease in autoantibodies, and a change of biomarkers. IA with Miltenyi's TheraSorb® column will be performed in the approved use. Patients who have symptom improvement after the 1st IA will receive two additional IAs at 3 and 6 months, which will also be documented. Symptom severity will be assessed by online questionnaires and at repeated time points.

Patients will be recruited for IA from the investigators' ongoing observational study with a follow-up of at least six months without disease improvement (Kedor et al., 2022). Patients have received a comprehensive diagnostic assessment to exclude other diseases, central nervous system, or organ comorbidity. ß2R autoantibodies in serum are determined by ELISA (Celltrend). Within four weeks prior to IA, patients will be assessed for eligibility for study participation by clinical investigation, laboratory analysis, and symptom questionnaires. The first ten patients will be treated end of August - mid of October and analyzed for efficacy until the beginning of December 2022 with a grant from the Weidenhammer-Zoebele foundation. The subsequent ten patients will be treated and analyzed with funding from the Federal Ministry of Education and Research(BMBF). These ten patients will also receive vessel diagnostics before (within four weeks) and four weeks after the first IA. In all 20 patients, blood will be collected the week before and four weeks after the first IA. All visits and treatments will take place in outpatient clinics.

Antibody depletion in PCS using IA has yet to be investigated in a clinical trial. The results of this observational study will provide the basis for a RCT using IA and, in responders, consecutive B-cell depleting therapy with an anti-CD20 monoclonal antibody versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients aged 18-65 years with a diagnosis of Post-COVID ME/CFS according to the Canadian Consensus Criteria (CCC) or fulfilling CCC with exertion intolerance with symptom worsening (post exertional malaise = PEM) duration of less than 14 hours (thus fulfilling Institute of Medicine criteria)
* Evidence of COVID infection at disease onset (PCR) or N-IgG
* Detection of autoantibodies (elevated ß2 receptor adrenergic autoantibodies)
* Immunoadsorption with the TheraSorb® column for 5 days
* Health insurance

Exclusion Criteria:

* Lack of willingness to store pseudonymized disease data as part of the study
* Pregnancy
* Other illnesses that do not allow the diagnosis of PCS to be made with certainty (e.g., heart failure, lung disease, severe depression, cancer)
* Acute infection (COVID, HIV, hepatitis)
* Severe fatigue disease with bedriddenness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the investigators' outpatient clinic who meet the CCC for ME/CFS (PEM for at least 14h or longer) and who are found to have elevated ß2R autoantibodies will be offered an IA and participation in this observational study. Also, PCS patients who do not meet CCC criteria due to shorter PEM (< 14h) but meet Systemic Exertion Intolerance Disease criteria may receive IA and be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | 4 weeks after first IA
  The Short Form 36 Health Survey (SF-36) is an established and widely used health-related quality of life measure. The Physical Function (PF) domain asks patients to report limitations on ten mobility activities, such as walking specified distances, carrying groceries, and bathing or dressing. Scores are weighted and transformed into a scale ranging from 0 (greatest possible health restrictions, i.e., severe disability) to 100 (no health restrictions). An intra-patient change of 10 points in SF-36-PF from baseline to week four is considered clinically meaningful.

SECONDARY OUTCOMES:
Efficacy of repeat immunoadsorptions (IA) on Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | 3 - 6 months after first IA
  Patients who have meaningful improvements in PF after the first IA, will receive two additional IAs at 3 and 6 months. Enhanced efficacy of repeat IAs on PF as measured by the SF-36 will be documented and assessed.
Response duration of repeat immunoadsorptions (IA) on Physical Function (PF) as measured by the Short Form 36 Health Survey Questionnaire (SF-36) | 3 - 6 months after first IA
  Additive effect of repeat IA to increase response duration after each IA cycle. Response duration assessed by SF-36 PF (> 10 points).
Improvement in ability to work in daily hours | 12 months after last IA
  Number of patients with an intra-patient change in his/her/their ability to work in daily hours from 6 months before first IA to 12 months after last IA.
Improvement in physical and mental fatigue as measured by the Chalder Fatigue Scale | 4 weeks after first IA; 6 and 12 months after last IA
  The Chalder Fatigue Scale measures the extent and severity of tiredness and has been used in multiple randomized trials of behavioral interventions in patients with ME/CFS. Each of the 11 items is answered on a 4-point scale with an overall score ranging from 0 (asymptomatic) to 33 (maximum symptomology). Intra-patient change in physical and mental fatigue from baseline to follow-up points will be documented as indexed by the Chalder Fatigue Scale.
Improvement in fatigue as measured by the Fatigue Severity Score (FSS) | 4 weeks after first IA; 6 and 12 months after last IA
  The Fatigue Severity Scale (FSS) is a 9-item scale that measures the severity of fatigue and its effect on a person's activities and lifestyle. Answers are scored on a seven-point scale (1 = strongly disagree; 7 = strongly agree). Thus, the minimum score is 9 (no fatigue), and the highest is 63 (heavy fatigue). Intra-patient change in fatigue severity from baseline to follow-up points will be documented as indexed by the FSS.
Improvement in symptoms of myalgic encephalomyelitis (ME)/ chronic fatigue syndrome (CFS) as measured by Canadian Consensus Criteria (CCC) Symptom Score | 4 weeks after first IA; 6 and 12 months after last IA
  The Canadian Consensus Criteria (CCC) Symptom Score quantifies ME/CFS symptoms. Its score ranges from 1 (no symptoms) to 10 (extreme symptoms). Intra-patient change in ME/CFS symptoms from baseline to follow-up points will be documented as indexed by the CCC Symptom Score.
Improvement in symptoms of autonomic dysfunction as measured by the Composite Autonomic Symptom Score (COMPASS-31) | 4 weeks after first IA; 6 and 12 months after last IA
  The Composite Autonomic Symptom Score (COMPASS-31) is a refined, internally consistent, and markedly abbreviated quantitative measure of autonomic symptoms. It is based on the original Autonomic Symptom Profile (ASP) and COMPASS, applies a much-simplified scoring algorithm, and is suitable for widespread use in autonomic research and practice. It evaluates six domains of autonomic function: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor domains. The score ranges from 0 (no symptoms) to 100 (strong autonomic dysfunction). Intra-patient change in autonomic dysfunction from baseline to follow-up points will be documented as indexed by the COMPASS-31.
Improvement in hand grip strength | 4 weeks after first IA; 6 and 12 months after last IA
  Intra-patient change in hand grip strength from baseline to follow-up points assessed using the Handgrip-Muscle-Fatigue Test
Improvement of vascular regulation as indexed by the reactive hyperemia index (RHI) assessed using Endopat. | 6 and 12 months after last IA
  Intra-patient change in endothelial cell function from baseline to follow-up points assessed using Endopat
Improvement in symptoms of orthostatic intolerance assessed using the Passive Standing Test | 4 weeks after first IA; 6 and 12 months after last IA
  Intra-patient change in orthostatic intolerance from baseline to follow-up points assessed using the Passive Standing Test.
Decrease in ß2R autoantibodies and soluble biomarkers of disease | 4 weeks after first IA; 6 and 12 months after last IA
  Intra-patient change in ß2R autoantibodies and soluble biomarkers of disease from baseline to follow-up points assessed
Verification of tolerability | 4 weeks after last IA
  Number of patients tolerating the IA treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kedor C, Freitag H, Meyer-Arndt L, Wittke K, Hanitsch LG, Zoller T, Steinbeis F, Haffke M, Rudolf G, Heidecker B, Bobbert T, Spranger J, Volk HD, Skurk C, Konietschke F, Paul F, Behrends U, Bellmann-Strobl J, Scheibenbogen C. A prospective observational study of post-COVID-19 chronic fatigue syndrome following the first pandemic wave in Germany and biomarkers associated with symptom severity. Nat Commun. 2022 Aug 30;13(1):5104. doi: 10.1038/s41467-022-32507-6. PMID 36042189
- [Background] Sotzny F, Blanco J, Capelli E, Castro-Marrero J, Steiner S, Murovska M, Scheibenbogen C; European Network on ME/CFS (EUROMENE). Myalgic Encephalomyelitis/Chronic Fatigue Syndrome - Evidence for an autoimmune disease. Autoimmun Rev. 2018 Jun;17(6):601-609. doi: 10.1016/j.autrev.2018.01.009. Epub 2018 Apr 7. PMID 29635081
- [Background] Freitag H, Szklarski M, Lorenz S, Sotzny F, Bauer S, Philippe A, Kedor C, Grabowski P, Lange T, Riemekasten G, Heidecke H, Scheibenbogen C. Autoantibodies to Vasoregulative G-Protein-Coupled Receptors Correlate with Symptom Severity, Autonomic Dysfunction and Disability in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. J Clin Med. 2021 Aug 19;10(16):3675. doi: 10.3390/jcm10163675. PMID 34441971
- [Background] Scheibenbogen C, Loebel M, Freitag H, Krueger A, Bauer S, Antelmann M, Doehner W, Scherbakov N, Heidecke H, Reinke P, Volk HD, Grabowski P. Immunoadsorption to remove ss2 adrenergic receptor antibodies in Chronic Fatigue Syndrome CFS/ME. PLoS One. 2018 Mar 15;13(3):e0193672. doi: 10.1371/journal.pone.0193672. eCollection 2018. PMID 29543914
- [Background] Tolle M, Freitag H, Antelmann M, Hartwig J, Schuchardt M, van der Giet M, Eckardt KU, Grabowski P, Scheibenbogen C. Myalgic Encephalomyelitis/Chronic Fatigue Syndrome: Efficacy of Repeat Immunoadsorption. J Clin Med. 2020 Jul 30;9(8):2443. doi: 10.3390/jcm9082443. PMID 32751659
- [Derived] Stein E, Heindrich C, Wittke K, Kedor C, Kim L, Freitag H, Kruger A, Tolle M, Scheibenbogen C. Observational Study of Repeat Immunoadsorption (RIA) in Post-COVID ME/CFS Patients with Elevated ss2-Adrenergic Receptor Autoantibodies-An Interim Report. J Clin Med. 2023 Oct 9;12(19):6428. doi: 10.3390/jcm12196428. PMID 37835071